CLINICAL TRIAL: NCT02607956
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of GS-9883/Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study to Evaluate the Safety and Efficacy of Bictegravir/Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Alafenamide in Human Immunodeficiency Virus (HIV-1) Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-380-1490; 2015-003988-10 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: HIV-1 Infection
Keywords: HIV
MeSH Terms: interventions — dolutegravir; emtricitabine tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- B/F/TAF (Experimental): B/F/TAF + DTG + F/TAF placebo administered without regard to food for at least 144 weeks.
  Interventions: Drug: B/F/TAF; Drug: DTG Placebo; Drug: F/TAF Placebo
- DTG + F/TAF (Active Comparator): DTG + F/TAF+ B/F/TAF placebo administered without regard to food for at least 144 weeks.
  Interventions: Drug: DTG; Drug: F/TAF; Drug: B/F/TAF Placebo
- Open-label Phase B/F/TAF from B/F/TAF (Experimental): After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF
- Open-label Phase B/F/TAF from DTG + F/TAF (Experimental): After Week 144, participants will continue to take their blinded study drug and attend visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants will be given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF is not commercially available will be given the option to continue OL B/F/TAF until the product becomes accessible through an access program or until Gilead elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: DTG — 50 mg tablets administered orally, once daily
  Other Names: Tivicay®
  Arms: DTG + F/TAF
Drug: F/TAF — 200/25 mg tablets administered orally, once daily
  Other Names: Descovy®
  Arms: DTG + F/TAF
Drug: B/F/TAF — 50/200/25 milligrams (mg) FDC tablets administered orally, once daily
  Other Names: GS-9883/F/TAF; Biktarvy®
  Arms: B/F/TAF; Open-label Phase B/F/TAF from B/F/TAF; Open-label Phase B/F/TAF from DTG + F/TAF
Drug: DTG Placebo — Tablets administered orally, once daily
  Arms: B/F/TAF
Drug: F/TAF Placebo — Tablets administered orally, once daily
  Arms: B/F/TAF
Drug: B/F/TAF Placebo — Tablets administered orally, once daily
  Arms: DTG + F/TAF

SUMMARY:
This primary objective of this study is to evaluate the efficacy of a fixed dose combination (FDC) containing bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus dolutegravir (DTG) + a FDC containing emtricitabine/tenofovir alafenamide (F/TAF) in HIV-1 infected, antiretroviral treatment-naive adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Antiretroviral treatment naive (≤ 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection) except the use for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), up to one month prior to screening
* Plasma HIV-1 ribonucleic acid (RNA) levels ≥ 500 copies per milliliter (mL) at screening
* Adequate renal function: Estimated glomerular filtration rate ≥ 30 mL per minute (min) (≥ 0.50 mL per second (sec)) according to the Cockcroft-Gault formula

Key Exclusion Criteria:

* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening
* Decompensated cirrhosis (eg, ascites, encephalopathy, or variceal bleeding)
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* Females who are pregnant (as confirmed by positive serum pregnancy test)
* Females who are breastfeeding

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2021-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (97):
- United States (58):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Sacramento, California
  - Optimus Medical - ClinEdge - PPDS, San Francisco, California
  - Kaiser Permanente, San Leandro, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Oakland Park, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Newark, New Jersey
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cone Health Regional Center for Infectious Disease, Greensboro, North Carolina
  - Greenville, North Carolina
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Bellaire, Texas
  - Dallas, Texas
  - AIDS Arms Inc, Dallas, Texas
  - North Texas Infectious Diseases Consultants PA, Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Australia (6):
  - Sydney, New South Wales
  - Carlton, Victoria
  - Clayton, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
  - Prahran Market Clinic, Prahran, Victoria
- Belgium (2):
  - Antwerp
  - Ghent
- Canada (5):
  - McGill University Health Center, Montreal
  - Ottawa
  - Sunnybrook Health Sciences Centre, Toronto
  - Toronto
  - Winnipeg
- Santo Domingo, Dominican Republic
- France (3):
  - Montpellier
  - CHU de Nice Archet I, Nice
  - Tourcoing
- Germany (7):
  - Berlin
  - Uniklinik Köln, Cologne
  - Düsseldorf
  - Essen
  - Frankfurt
  - Hamburg
  - München
- Italy (3):
  - Bergamo
  - Milan
  - Roma
- San Juan, Puerto Rico
- Spain (6):
  - Alicante
  - Badalona
  - Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Málaga
  - Vigo
- United Kingdom (5):
  - Birmingham
  - London
  - Chelsea and Westminster NHS Trust, London
  - St George's Healthcare NHS Trust, London
  - Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Sax PE, Pozniak A, Montes ML, Koenig E, DeJesus E, Stellbrink HJ, Antinori A, Workowski K, Slim J, Reynes J, Garner W, Custodio J, White K, SenGupta D, Cheng A, Quirk E. Coformulated bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection (GS-US-380-1490): a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2073-2082. doi: 10.1016/S0140-6736(17)32340-1. Epub 2017 Aug 31. PMID 28867499
- [Result] Gupta SK, Post FA, Arribas JR, Eron JJ Jr, Wohl DA, Clarke AE, Sax PE, Stellbrink HJ, Esser S, Pozniak AL, Podzamczer D, Waters L, Orkin C, Rockstroh JK, Mudrikova T, Negredo E, Elion RA, Guo S, Zhong L, Carter C, Martin H, Brainard D, SenGupta D, Das M. Renal safety of tenofovir alafenamide vs. tenofovir disoproxil fumarate: a pooled analysis of 26 clinical trials. AIDS. 2019 Jul 15;33(9):1455-1465. doi: 10.1097/QAD.0000000000002223. PMID 30932951
- [Result] Stellbrink HJ, Arribas JR, Stephens JL, Albrecht H, Sax PE, Maggiolo F, Creticos C, Martorell CT, Wei X, Acosta R, Collins SE, Brainard D, Martin H. Co-formulated bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir with emtricitabine and tenofovir alafenamide for initial treatment of HIV-1 infection: week 96 results from a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet HIV. 2019 Jun;6(6):e364-e372. doi: 10.1016/S2352-3018(19)30080-3. Epub 2019 May 5. PMID 31068272
- [Result] Acosta RK, Willkom M, Martin R, Chang S, Wei X, Garner W, Lutz J, Majeed S, SenGupta D, Martin H, Quirk E, White KL. Resistance Analysis of Bictegravir-Emtricitabine-Tenofovir Alafenamide in HIV-1 Treatment-Naive Patients through 48 Weeks. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e02533-18. doi: 10.1128/AAC.02533-18. Print 2019 May. PMID 30803969
- [Result] Acosta R, Willkom M, Martin R, Chang S, Liu X, Hedskog C, et al. Low-frequency resistance variants in ART-naive participants do not affect bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) triple therapy outcome. [Poster MOPEB242]. 10th IAS Conference on HIV Science (IAS 2019); 2019 July 21-24; Mexico City, Mexico.
- [Result] Johnson M, Taylor S, Wei X, Collins SE, Martin H. Hepatic Safety of Bictegravir/Emtricitabine/Tenofovir Alafenamide [Poster P061]. 25th Annual Conference of the British HIV Association; 2019 02-05 April; Bournemouth, United Kingdom.
- [Result] Gupta S, Mills A, Brinson C, Workowski K, Clarke A, Antinori A, et al. 96 Week Efficacy and Safety of B/F/TAF in Treatment-Naïve Adults and Adults ≥50 Years [Poster 502]. CROI 2019; 2019 04-07 March; Seattle, WA.
- [Result] Acosta R, White K, Garner W, Wei X, Andreatta K, Willkom M, et al. HIV-1 subtype (B or non-B) had no impact on the efficacy of B/F/TAF or resistance development in five phase 3 treatment-naïve or switch studies. [Poster THPEB077]. 22nd International AIDS Conference; 2018 July 23-27; Amsterdam, Netherlands.
- [Result] White K, Kulkarni R, Willkom M, Martin R, Chang S, Wei X, et al. Pooled week 48 efficacy and baseline resistance: B/F/TAF in treatment-naive patients. [Poster 532]. Conference on Retroviruses and Opportunistic Infections; 2018 March 4-7; Boston, USA.
- [Result] Wohl D, Clarke A, Maggiolo F, Garner W, Laouri M, Martin H, Quirk E. Patient-Reported Symptoms Over 48 Weeks Among Participants in Randomized, Double-Blind, Phase III Non-inferiority Trials of Adults with HIV on Co-formulated Bictegravir, Emtricitabine, and Tenofovir Alafenamide versus Co-formulated Abacavir, Dolutegravir, and Lamivudine. Patient. 2018 Oct;11(5):561-573. doi: 10.1007/s40271-018-0322-8. PMID 29956087
- [Result] Wohl DA, Yazdanpanah Y, Baumgarten A, Clarke A, Thompson MA, Brinson C, Hagins D, Ramgopal MN, Antinori A, Wei X, Acosta R, Collins SE, Brainard D, Martin H. Bictegravir combined with emtricitabine and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection: week 96 results from a randomised, double-blind, multicentre, phase 3, non-inferiority trial. Lancet HIV. 2019 Jun;6(6):e355-e363. doi: 10.1016/S2352-3018(19)30077-3. Epub 2019 May 5. PMID 31068270
- [Result] Acosta R, Andreatta K, D'Antoni M, Collins S, Martin H, White K. HIV Viral Blips in Adults Treated with INSTI-Based Regimens Through 144 Weeks. [Poster 540]. Conference on Retroviruses and Opportunistic Infections 2020 (CROI 2020); 2020 March 8-11; Boston, Massachusetts.
- [Result] Mills A, Gupta SK, Brinson C, Workowski K, Clarke A, Antinori A, Stephens JL, et al. 144-Week Efficacy and Safety of B/F/TAF in Treatment-Naive Adults Age ≥50 Years. [Poster 477]. Conference on Retroviruses and Opportunistic Infections 2020 (CROI 2020); 2020 March 8-11; Boston, Massachusetts.
- [Result] Orkin C, DeJesus E, Sax PE, Arribas JR, Gupta SK, Martorell C, Stephens JL, Stellbrink HJ, Wohl D, Maggiolo F, Thompson MA, Podzamczer D, Hagins D, Flamm JA, Brinson C, Clarke A, Huang H, Acosta R, Brainard DM, Collins SE, Martin H; GS-US-380-1489; GS-US-380-1490 study investigators. Fixed-dose combination bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir-containing regimens for initial treatment of HIV-1 infection: week 144 results from two randomised, double-blind, multicentre, phase 3, non-inferiority trials. Lancet HIV. 2020 Jun;7(6):e389-e400. doi: 10.1016/S2352-3018(20)30099-0. PMID 32504574
- [Result] Ramgopal M, Maggiolo F, Ward D, Leboucche B, Rizzardini G, Molina JM, et al. Pooled Analysis of 4 International Trials of Bictegravir/Emtrictabine/Tenofovir Alafenamide (B/F/TAF) in Adults Aged ≥ 65 Years Demonstrating Safety and Efficacy: Week 48 Results. [Oral OAB0403].AIDS 2020; 2020 July 6-10; Virtual.
- [Result] Acosta R, Andreatta K, D'Antoni M, Collins S, Martin H, White K. Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) shows high efficacy in clinical study participants infected with HIV-1 subtype F. [Poster P124]. HIV Drug Therapy 2020 (HIV Glasgow 2020); 2020 October 5-8; Glasgow, United Kingdom.
- [Result] Acosta R, Chen G, Chang S, Martin R, Wang X, Huang H, et al. HIV with Transmitted Drug Resistance Is Durably Suppressed by B/F/TAF at Week 144. [Poster 430]. Conference on Retroviruses and Opportunistic Infections 2021 (CROI 2021); 2021 June 3-November 3; Virtual.
- [Result] Acosta RK, Chen GQ, Chang S, Martin R, Wang X, Huang H, Brainard D, Collins SE, Martin H, White KL. Three-year study of pre-existing drug resistance substitutions and efficacy of bictegravir/emtricitabine/tenofovir alafenamide in HIV-1 treatment-naive participants. J Antimicrob Chemother. 2021 Jul 15;76(8):2153-2157. doi: 10.1093/jac/dkab115. PMID 33880558
- [Result] Workowski K, Orkin C, Sax P, Hagins D, Koenig E, Stephens JL, et al. Four-Year Outcomes of B/F/TAF in Treatment-Naïve Adults [Poster 415]. Conference on Retroviruses and Opportunistic Infections 2021 (CROI 2021); 2021 June 3-November 3; Virtual.
- [Result] Acosta R, Chen G, Qin L, Wang X, Huang H, Hindman J, et al. Achievement of Undetectable HIV-1 RNA in the B/F/TAF Treatment-Naive Clinical Trials. [Poster PEB150]. 11th IAS Conference on HIV Science (IAS 2021); 2021 July 18-21; Virtual.
- [Result] Acosta R, Chen G, Huang H, Liu H, White K. Unreturned Pill Bottles in the 1489 and 1490 Clinical Trials: An Important Measure of Poor Adherence That Is Often Ignored in Pill Count Calculations. [Poster 902]. IDWeek 2021; 2021 September 29-October 3; Virtual.
- [Result] Arribas J, Orkin C, Maggiolo F, Antinori A, Lazzarin A, Yasdanpanah, et al. Long-term Analysis of B/F/TAF in Treatment-Naïve Adults Living With HIV Through Four Years of Follow-up. [PEB151]. 11th IAS Conference on HIV Science (IAS 2021); 2021 July 18-21; Virtual.
- [Result] Daar E, Orkin C, Sax P, Stephens J, Koenig E, Clarke A, et al. Incidence of Metabolic Complications Among Treatment-naïve Adults Living With HIV-1 Randomized to B/F/TAF, DTG/ABC/3TC or DTG+F/TAF After 3 Years. [Oral 69]. IDWeek 2021; 2021 September 29- October 3; Virtual.
- [Result] Pozniak A, et al. Outcomes 48 Weeks After Switching From DTG/ABC/3TC or DTG+F/TAF to B/F/TAF. [PE2/68]. 18th European AIDS Conference (EAC 2021), 2021 October 27-30; London, United Kingdom.
- [Derived] Sax PE, Hindman JT, Martin H, Wohl D. Two 5-year studies of bictegravir/emtricitabine/tenofovir alafenamide in people with HIV: a plain-language summary. Future Microbiol. 2024;19(14):1185-1193. doi: 10.1080/17460913.2024.2372231. Epub 2024 Sep 4. PMID 39229805
- [Derived] Orkin C, Antinori A, Rockstroh JK, Moreno-Guillen S, Martorell CT, Molina JM, Lazzarin A, Maggiolo F, Yazdanpanah Y, Andreatta K, Huang H, Hindman JT, Martin H, Pozniak A. Switch to bictegravir/emtricitabine/tenofovir alafenamide from dolutegravir-based therapy. AIDS. 2024 Jun 1;38(7):983-991. doi: 10.1097/QAD.0000000000003865. Epub 2024 Feb 21. PMID 38349226
- [Derived] Sax PE, Arribas JR, Orkin C, Lazzarin A, Pozniak A, DeJesus E, Maggiolo F, Stellbrink HJ, Yazdanpanah Y, Acosta R, Huang H, Hindman JT, Martin H, Baeten JM, Wohl D; GS-US-380-1489 and GS-US-380-1490 study investigators. Bictegravir/emtricitabine/tenofovir alafenamide as initial treatment for HIV-1: five-year follow-up from two randomized trials. EClinicalMedicine. 2023 May 11;59:101991. doi: 10.1016/j.eclinm.2023.101991. eCollection 2023 May. PMID 37200995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at centers in Australia, Europe, North America, and the Dominican Republic. The first participant was screened on 11 November 2015. The last study visit occurred on 05 July 2021.
Pre-assignment Details: 742 participants were screened.
Groups:
- B/F/TAF: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) tablets fixed-dose combination (FDC) + dolutegravir (DTG) placebo + F/TAF placebo orally once daily for at least 144 weeks without regard to food.
- DTG + F/TAF: DTG (50 mg) + F/TAF (200/25 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks without regard to food.
- B/F/TAF to B/F/TAF; DTG + F/TAF to B/F/TAF: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive open-label (OL) B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Period: Double-Blinded Phase
Arm/Group | B/F/TAF | DTG + F/TAF | B/F/TAF to B/F/TAF | DTG + F/TAF to B/F/TAF
Started | 327 | 330 | 0 | 0
Completed | 266 | 277 | 0 | 0
Not Completed | 61 | 53 | 0 | 0
Not completed — Withdrew Consent | 17 | 19 | 0 | 0
Not completed — Lost to Follow-up | 19 | 16 | 0 | 0
Not completed — Randomized but never treated | 7 | 5 | 0 | 0
Not completed — Investigator's Discretion | 7 | 2 | 0 | 0
Not completed — Death | 4 | 4 | 0 | 0
Not completed — Adverse Event | 4 | 3 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 0
Not completed — Non-Compliance with Study Drug | 0 | 3 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | B/F/TAF | DTG + F/TAF | B/F/TAF to B/F/TAF | DTG + F/TAF to B/F/TAF
Started | 0 (At the End of Blinded Treatment Visit, participants were given the option to receive B/F/TAF FDC in an OL extension phase for up to 96 weeks.) | 0 (At the End of Blinded Treatment Visit, participants were given the option to receive B/F/TAF FDC in an OL extension phase for up to 96 weeks.) | 254 (66 participants from the Double-Blinded Phase did not enter the Open-Label Extension Phase.) | 265 (60 participants from the Double-Blinded Phase did not enter the Open-Label Extension Phase.)
Completed | 0 | 0 | 225 | 235
Not Completed | 0 | 0 | 29 | 30
Not completed — Withdrew Consent | 0 | 0 | 10 | 16
Not completed — Lost to Follow-up | 0 | 0 | 14 | 6
Not completed — Death | 0 | 0 | 1 | 3
Not completed — Investigator's Discretion | 0 | 0 | 2 | 2
Not completed — Non Compliance with Study Drug | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were randomized into the study and received at least 1 dose of the study drug.
Groups:
- B/F/TAF: Blinded Phase: B/F/TAF (50/200/25 mg) FDC + DTG placebo + F/TAF placebo orally once daily for at least 144 weeks, without regard to food
  Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
- DTG + F/TAF: Blinded Phase: DTG (50 mg) + F/TAF (200/25 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks, without regard to food
  Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | DTG + F/TAF | Total
Number analyzed (Participants) | 320 | 325 | 645
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12.3) | 37 (11.6) | 37 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 280 | 288 | 568
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 10 | 17
  Black | 97 | 100 | 197
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 183 | 195 | 378
  Other | 31 | 19 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 81 | 164
  Not Hispanic or Latino | 237 | 244 | 481
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12 | 9 | 21
  Belgium | 4 | 4 | 8
  United States | 193 | 193 | 386
  Dominican Republic | 27 | 18 | 45
  Italy | 15 | 18 | 33
  United Kingdom | 21 | 23 | 44
  Australia | 4 | 10 | 14
  France | 7 | 5 | 12
  Germany | 20 | 28 | 48
  Spain | 17 | 17 | 34
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.39 (0.730) | 4.42 (0.669) | 4.41 (0.700)
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 254 | 271 | 525
  > 100,000 ≤ 400,000 copies/mL | 54 | 41 | 95
  > 400,000 copies/mL | 12 | 13 | 25
CD4 Cell Count [Mean (Standard Deviation); unit: Cells/µL] | 457 (255.3) | 454 (231.5) | 456 (243.4)
CD4 Cell Count Categories [Count of Participants; unit: Participants]
  < 50 cells/μL | 15 | 13 | 28
  ≥ 50 to < 200 cells/μL | 29 | 21 | 50
  ≥ 200 to < 350 cells/μL | 67 | 77 | 144
  ≥ 350 to < 500 cells/μL | 91 | 94 | 185
  ≥ 500 cells/μL | 118 | 120 | 238

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- B/F/TAF: Blinded Phase: B/F/TAF (50/200/25 mg) FDC + DTG placebo + F/TAF placebo orally once daily for at least 144 weeks, without regard to food.
- DTG + F/TAF: Blinded Phase: DTG (50 mg) + F/TAF (200/25 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 144 weeks, without regard to food.
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 89.4 | 92.9
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Non-Inferiority — A sample of approximately 600 participants randomized 1:1 achieves at least 95% power using a non-inferiority margin of 12% assuming a response rate in both groups of 91% (Reference Genvoya studies) and a one-sided alpha level of 0.025; Difference in Percentages = -3.5, 95.002% CI 2-sided [-7.9 to 1.0] — Differences in percentages of participants between groups and their 95.002% CIs were calculated based on Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Superiority; p = 0.12, Cochran-Mantel-Haenszel; p-value was calculated from CMH test stratified by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)

2. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 84.1 | 86.5
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-7.9 to 3.2] — Differences in percentages of participants between groups and their 95% CIs were calculated based on MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.41, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 144 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 144 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 144
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 81.9 | 84.0
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; Difference in Percentages = -1.9, 95% CI 2-sided [-7.8 to 3.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.52, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 82.2 | 87.1
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; Difference in Percentages = -3.9, 95% CI 2-sided [-9.4 to 1.5] — The differences in percentages of participants between treatment groups and their 95% CIs were calculated based on the MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) and region stratum (US vs. Ex-US)
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.16, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

5. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 96 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 77.5 | 80.3
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; Difference in Percentages = -2.5, 95% CI 2-sided [-8.8 to 3.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.44, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 20 Copies/mL at Week 144 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 144 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 144
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 320 | 325
percentage of participants | 77.5 | 79.1
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; Difference in Percentages = -1.1, 95% CI 2-sided [-7.4 to 5.3] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.74, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 294 | 308
log10 copies/mL | -3.07 (0.719) | -3.12 (0.672)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.081, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = 0.08, 95% CI 2-sided [-0.01 to 0.17] — Difference in least-squares mean (LSM), and its 95% confidence interval (CI) were adjusted by baseline HIV-1 RNA stratum and region stratum

8. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 276 | 291
log10 copies/mL | -3.08 (0.703) | -3.10 (0.713)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.18, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = 0.06, 95% CI 2-sided [-0.03 to 0.15] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

9. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 270 | 280
log10 copies/mL | -3.06 (0.731) | -3.11 (0.672)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.054, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = 0.09, 95% CI 2-sided [0.00 to 0.18] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 290 | 304
cells/μL | 180 (166.2) | 201 (165.9)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.096, ANOVA; P-value was adjusted by the baseline HIV-1 RNA and region stratum; Difference in LSM = -23, 95% CI 2-sided [-49 to 4] — Difference in LSM, and its 95% CI were adjusted by the baseline HIV-1 RNA and region stratum

11. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 269 | 285
cells/μL | 237 (204.2) | 281 (209.3)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.008, ANOVA; P-value was adjusted by the baseline HIV-1 RNA and region stratum; Difference in LSM = -47, 95% CI 2-sided [-81 to -12] — Difference in LSM, and its 95% CI were adjusted by the baseline HIV-1 RNA and region stratum

12. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 144
Time Frame: Baseline, Week 144
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 262 | 277
cells/μL | 278 (236.6) | 289 (218.5)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Other; p = 0.48, ANOVA; p-value was adjusted by baseline HIV-1 RNA stratum and region stratum; Difference in LSM = -14, 95% CI 2-sided [-52 to 25] — Difference in LSM, and its 95% CI were adjusted by baseline HIV-1 RNA stratum and region stratum

13. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 Open-Label as Defined by Missing = Excluded Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL was analyzed using Missing = Excluded for imputing missing HIV-1 RNA values using the All B/F/TAF Analysis Set for the all B/F/TAF analysis. All missing data was excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation). The denominator for percentages at a visit was the number of participants in the all B/F/TAF analysis set with nonmissing HIV-1 RNA value at that visit.
Time Frame: Baseline, open-label Week 48
Population: Participants in All B/F/TAF Analysis Set (who were randomized into the randomized phase of the study and received at least 1 dose of the B/F/TAF in the randomized phase or at least 1 dose of the B/F/TAF in the open label extension phase) with available data were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Missing = Excluded analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All B/F/TAF: Blinded Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) tablets fixed-dose combination (FDC) + dolutegravir (DTG) placebo + F/TAF placebo orally once daily for at least 144 weeks without regard to food.
  Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
- DTG + F/TAF to B/F/TAF: Open Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 243 | 225
percentage of participants | 99.2 [97.1 to 99.9] | 99.6 [97.5 to 100.0]

14. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 48 Open-Label as Defined by Missing = Failure Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL was analyzed using Missing = Failure for imputing missing HIV-1 RNA values using the All B/F/TAF Analysis Set for the all B/F/TAF analysis. All missing data was treated as HIV-1 RNA ≥ 50 copies/mL. The denominator for percentages was the number of participants in all B/F/TAF analysis set.
Time Frame: Baseline, open-label Week 48
Population: Participants in the All B/F/TAF Analysis Set were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Missing = Failure analysis, it included all participants from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 320 | 265
percentage of participants | 75.3 [70.2 to 79.9] | 84.5 [79.6 to 88.7]

15. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 Open-Label as Defined by Missing = Excluded Algorithm
Description: as for outcome 13
Time Frame: Baseline, open-label Week 96
Population: Participants in All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Missing = Excluded analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DTG + F/TAF to B/F/TAF: Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 219 | 234
percentage of participants | 99.5 [97.5 to 100.0] | 99.1 [96.9 to 99.9]

16. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA < 50 Copies/mL at Week 96 Open-Label as Defined by Missing = Failure Algorithm
Description: as for outcome 14
Time Frame: Baseline, open-label Week 96
Population: Participants in the All B/F/TAF Analysis Set were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Missing = Failure analysis, it included all participants from the Randomized Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 320 | 265
percentage of participants | 68.1 [62.7 to 73.2] | 87.5 [83.0 to 91.3]

17. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48 Open-Label
Time Frame: Baseline, open-label Week 48
Population: Participants in the All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 48 open-label time point refers to Week 192; for Change from Baseline in CD4 Cell Count analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Mean (Standard Deviation); unit: cells/μL
Groups:
- All B/F/TAF: Blinded Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) tablets fixed-dose combination (FDC) + dolutegravir (DTG) placebo + F/TAF placebo orally once daily for at least 144 weeks without regard to food
  Open-Label Extension Phase: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 241 | 223
cells/μL | 304 (249.2) | 9 (198.0)

18. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96 Open-Label
Time Frame: Baseline, open-label Week 96
Population: Participants in the All B/F/TAF Analysis Set with available data were analyzed. For the B/F/TAF group, Week 96 open-label time point refers to Week 240; for Change from Baseline in CD4 Cell Count analysis, it included the available participants at that time point from the Randomized Phase.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | All B/F/TAF | DTG + F/TAF to B/F/TAF
Number analyzed (Participants) | 210 | 225
cells/µL | 336 (235.1) | -10 (181.1)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (maximum: 281.4 weeks) plus 30 days All-Cause Mortality: Randomization date through last visit/follow up date (maximum: 287.1 weeks)
Description: Adverse Events: Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
  All-Cause Mortality: All Randomized Analysis Set included all participants randomized into the study.
Groups:
- B/F/TAF to B/F/TAF; DTG + F/TAF to B/F/TAF: After Week 144, participants continued to take their blinded study drug and attended visits every 12 weeks until the End of Blinded Treatment Visit. Following the End of Blinded Treatment Visit, participants were given the option to receive OL B/F/TAF for 96 weeks. After the Week 96 OL Visit, participants in a country where B/F/TAF was not commercially available were given the option to continue OL B/F/TAF until the product became accessible through an access program or until Gilead elected to discontinue the study in that country, whichever occured first.
Arm/Group | B/F/TAF | DTG + F/TAF | B/F/TAF to B/F/TAF | DTG + F/TAF to B/F/TAF
All-Cause Mortality (participants affected / at risk) | 4/327 | 4/330 | 1/254 | 3/265
Serious Adverse Events (participants affected / at risk) | 64/320 | 46/325 | 20/254 | 32/265
Other Adverse Events (participants affected / at risk) | 250/320 | 262/325 | 165/254 | 163/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=320) | DTG + F/TAF (N=325) | B/F/TAF to B/F/TAF (N=254) | DTG + F/TAF to B/F/TAF (N=265)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Death (General disorders) | 0 | 2 | 1 | 2
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Amoebic dysentery (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 3 | 0 | 0 | 0
Anal infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 3 | 2 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Blister infected (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 6 | 1 | 1 | 2
Covid-19 (Infections and infestations) | 0 | 0 | 2 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection syphilitic (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 2 | 2
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 2 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rectal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Seasonal affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance use disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 2 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=320) | DTG + F/TAF (N=325) | B/F/TAF to B/F/TAF (N=254) | DTG + F/TAF to B/F/TAF (N=265)
Lymphadenopathy (Blood and lymphatic system disorders) | 24 | 23 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 23 | 23 | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 16 | 13 | 5 | 2
Constipation (Gastrointestinal disorders) | 16 | 15 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 66 | 54 | 15 | 15
Dyspepsia (Gastrointestinal disorders) | 21 | 14 | 2 | 5
Nausea (Gastrointestinal disorders) | 31 | 43 | 8 | 11
Toothache (Gastrointestinal disorders) | 16 | 9 | 5 | 3
Vomiting (Gastrointestinal disorders) | 23 | 22 | 5 | 5
Fatigue (General disorders) | 29 | 37 | 4 | 13
Pyrexia (General disorders) | 21 | 31 | 6 | 9
Anal chlamydia infection (Infections and infestations) | 18 | 18 | 11 | 8
Bronchitis (Infections and infestations) | 15 | 28 | 10 | 7
Chlamydial infection (Infections and infestations) | 14 | 26 | 5 | 6
Covid-19 (Infections and infestations) | 0 | 0 | 26 | 31
Gastroenteritis (Infections and infestations) | 15 | 18 | 5 | 8
Gonorrhoea (Infections and infestations) | 18 | 24 | 2 | 4
Influenza (Infections and infestations) | 27 | 24 | 15 | 11
Nasopharyngitis (Infections and infestations) | 51 | 62 | 19 | 22
Pharyngitis (Infections and infestations) | 22 | 11 | 4 | 1
Proctitis gonococcal (Infections and infestations) | 12 | 17 | 3 | 8
Sinusitis (Infections and infestations) | 25 | 10 | 10 | 5
Syphilis (Infections and infestations) | 34 | 33 | 20 | 17
Upper respiratory tract infection (Infections and infestations) | 44 | 54 | 15 | 17
Urinary tract infection (Infections and infestations) | 19 | 14 | 3 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 33 | 16 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 44 | 18 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 11 | 8 | 13
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 11 | 1 | 6
Dizziness (Nervous system disorders) | 17 | 20 | 7 | 5
Headache (Nervous system disorders) | 57 | 59 | 16 | 19
Anxiety (Psychiatric disorders) | 16 | 26 | 9 | 9
Depression (Psychiatric disorders) | 21 | 26 | 9 | 9
Insomnia (Psychiatric disorders) | 29 | 25 | 8 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 30 | 16 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 19 | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 15 | 27 | 7 | 11
Hypertension (Vascular disorders) | 19 | 22 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (7):
  • Study Protocol: Original (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/Prot_004.pdf
  • Study Protocol: Amendment 1 (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/Prot_005.pdf
  • Study Protocol: Amendment 2 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/Prot_006.pdf
  • Study Protocol: Amendment 3 (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/Prot_008.pdf
  • Statistical Analysis Plan: Original (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/SAP_007.pdf
  • Statistical Analysis Plan: Amendment 1 (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/SAP_009.pdf
  • Statistical Analysis Plan: Final Analysis (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02607956/SAP_010.pdf